CLINICAL TRIAL: NCT07344584
Title: A Prospective Pilot Study to Evaluate Safety and Effectiveness of GP0122 and GP0124 for Correction of Lines and Wrinkles in the Cheek Area
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 43CASH2210
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Wrinkle Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GP0122 (Active Comparator): Participants will receive GP0122 in the cheek area at baseline with an optional touch-up session 1 month after the initial session.
  Interventions: Device: GP0122
- GP0124 (Active Comparator): Participants will receive GP0124 in the cheek area at baseline with an optional touch-up session 1 month after the initial session.
  Interventions: Device: GP0124

INTERVENTIONS:
Device: GP0122 — Injectable gel.
  Arms: GP0122
Device: GP0124 — Injectable gel.
  Arms: GP0124

SUMMARY:
The primary objective of the study is to evaluate the safety of GP0122 and GP0124 for the correction of lines and wrinkles in the cheek area.

ELIGIBILITY:
Inclusion Criteria: Adult males or non-pregnant, non-breastfeeding adult females.

1. Participants with a GCWS At Rest score of Moderate or Severe on EACH side of the face, or Participants with a CSQS-CL score of Moderate, Severe, or Very severe on EACH side of the face.
2. Intent to undergo treatment for correction of lines and wrinkles in the cheek region.
3. Willing to abstain from any other facial plastic, surgical or cosmetic procedures in the cheek area for the duration of the study (e.g., laser or chemical resurfacing, needling, facelift, lifting threads, radiofrequency etc.).

   Inclusion criteria 4-5 apply only to female participants of childbearing potential:
4. Agrees to use an acceptable form of effective birth control for the duration of the study and is willing to take a urine pregnancy test (UPT) at screening, baseline and prior to receiving any study treatment.
5. Negative UPT at the screening and baseline visits.

Exclusion Criteria:

1. Known/previous allergy or hypersensitivity.
2. Known/previous allergy or hypersensitivity to local anesthetics.
3. Previous facial surgery (e.g., facelift) in the treatment area that in the Treating Investigator´s opinion.
4. Any previous aesthetic procedures or implants in the treatment area.
5. Presence of any disease or lesions in the treatment area.
6. An underlying known disease, a surgical or medical condition that would expose the participant to undue risk.
7. Use of concomitant medication that have the potential to prolong bleeding times.
8. Presence of any condition or situation, which in the opinion of the Treating Investigator makes the subject unable to complete the study per protocol.
9. Women who are pregnant or breast feeding, or women of childbearing potential who are not practicing adequate contraception or planning to become pregnant during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-16 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With all Adverse Events (AEs) | From Day 1 up to last visit (Up to 12 months)
Number of Participants With Post-Treatment Responses as Assessed Using Subject Diary Data | From Day 1 up to Day 28
Participant's Pain Assessment Using Numeric Pain Scale (NPS) Immediately Post Treatment and 30 Minutes Post Treatment | Immediately and 30 minutes after each treatment

SECONDARY OUTCOMES:
Responder Rates Based on the Treating Investigator's Live Assessment of the GCWS at Rest at Months 3, 6, 9 and 12 | At Months 3, 6, 9 and 12
Responder Rates Based on the Treating Investigator's Live Assessment of the CSQS-CL at Rest at Months 3, 6, 9 and 12 | At Months 3, 6, 9 and 12

IPD SHARING:
Plan to Share IPD: No